CLINICAL TRIAL: NCT00062270
Title: Neoadjuvant Chemoradiotherapy (Gemcitabine/Cisplatin and Taxotere) With or Without Co-Administration of ZD 1839 (Iressa) for Stage IIIA (N2) and Selective Stage IIIB Non-Small Cell Lung Cancer: Phase I-II Study
Brief Title: Neoadjuvant Chemoradiotherapy With or Without Gefitinib in Treating Patients With Stage IIIA or Stage IIIB Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000304674; UAB-0162; UAB-F020730006; ZENECA-ZD1839US-0207; AVENTIS-GIA-12139
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Gefitinib; Gemcitabine; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: gefitinib
Drug: gemcitabine hydrochloride
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of the tumor. Combining chemotherapy and radiation therapy with gefitinib before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase I/II trial to compare the effectiveness of neoadjuvant chemoradiotherapy with or without gefitinib in treating patients who are undergoing surgery for stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: Phase I:

* Determine the tolerability and toxicity of gefitinib in combination with chest radiotherapy in patients with stage IIIA or stage IIIB non-small cell lung cancer.

Phase II:

* Compare the pathologic response (complete response and rate of downstaging) in patients treated with neoadjuvant chemoradiotherapy with vs without gefitinib.
* Compare the feasibility and toxicity profile of these regimens in these patients.
* Compare the resection rates, time to progression, and overall survival of patients treated with these regimens.
* Correlate the percent decline in the fludeoxyglucose F 18 standardized uptake value as measured by position emission tomography with pathologic response at resection, time to progression, and overall survival in patients treated with these regimens.

OUTLINE:

* Phase I: This is an open-label, nonrandomized study.

  * Induction: Patients receive cisplatin IV over 60 minutes on day 1 and gemcitabine IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for a total of 2 courses in the absence of disease progression or unacceptable toxicity.
  * Consolidation: Within 3-4 weeks after the completion of induction therapy, patients undergo radiotherapy once daily 5 days a week for 5 weeks and receive oral gefitinib once daily concurrently.

A cohort of 3-6 patients receives consolidation chemoradiotherapy. If 2 of 6 patients experience dose-limiting toxicity, gefitinib is deleted from consolidation therapy in phase II arm II.

* Surgery: Patients without disease progression after consolidation therapy undergo thoracotomy within 3-5 weeks after consolidation.
* Maintenance: Beginning 2-4 weeks after surgery, patients receive oral gefitinib once daily for 6 months in the absence of disease progression.

  * Phase II: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.
* Arm I: Patients receive induction and consolidation therapy (with the exception of gefitinib) as in phase I. Patients also receive docetaxel IV over 60 minutes concurrently with radiotherapy during consolidation. Patients undergo surgery as in phase I.
* Arm II: Patients receive therapy (including gefitinib) as in phase I. Patients also receive docetaxel IV over 60 minutes concurrently with radiotherapy during consolidation.

Patients are followed every 6-8 weeks for the first 12 months and then every 4-6 months thereafter.

PROJECTED ACCRUAL: A total of 43-80 patients (3-6 patients for phase I and 40-74 patients [20-37 per treatment arm] for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage IIIA (T1-3, N2)

    * Positive (pathological) ipsilateral mediastinal node
  * Selective stage IIIB meeting all of the following criteria:

    * No pleural/pericardial effusion or superior vena cava syndrome
    * T4 due to invasion of carina, trachea, or mediastinal structures
    * Mediastinal N3 nodes (without supraclavicular or cervical adenopathy)
* Proof of N2 or N3 status requires surgical staging of the mediastinum (mediastinoscopy, mediastinotomy, or exploration)
* Expression of epidermal growth factor receptor (at least 1+) by immunohistochemistry
* Measurable disease by contrast CT scan allowed
* No bronchoalveolar cell carcinoma
* No prior diagnosis of lung cancer

PATIENT CHARACTERISTICS:

Age

* 19 and over

Performance status

* ECOG 0-1 (0-2 if albumin is at least 0.85 times lower limit of normal and weight loss within 3 months before diagnosis is no greater than 10%)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin normal
* AST and ALT no greater than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN

  * Alkaline phosphatase between 1.5-2 times ULN requires a negative bone scan for metastatic bone disease

Renal

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiac

* No myocardial infarction within the past 3 months
* No active angina
* No unstable heart rhythms
* No congestive heart failure

Pulmonary

* Post-resection predicted FEV_1% greater than 35%

  * Predicted FEV_1% is defined as FEV_1% times percent perfusion to uninvolved lung from quantitative lung V/Q scan report

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 weeks after study treatment
* No other uncontrolled medical illness
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No grade 2 or greater peripheral neuropathy
* No concurrent ocular inflammation or infection
* No prior severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No known severe hypersensitivity reaction to gefitinib or any of its excipients
* No prior severe allergic reaction to platinum-containing compounds or mannitol

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF]) during chemotherapy

Chemotherapy

* No prior chemotherapy for lung cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for lung cancer

Surgery

* Recovered from prior major surgery
* No concurrent ophthalmic surgery

Other

* More than 30 days since prior unapproved or investigational drugs
* No concurrent use of the following drugs:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Hypericum perforatum (St. John's Wort)
  * Warfarin
* No concurrent retinoids

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Determine the tolerability and toxicity of gefitinib in combination with chest radiotherapy in patients with stage IIIA or stage IIIB non-small cell lung cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, FACP, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States